CLINICAL TRIAL: NCT01453998
Title: Safety and Immunogenicity of a Booster Dose of New Formulations of GlaxoSmithKline Biologicals' DTPa-HBV-IPV/Hib Vaccine (GSK217744)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114843; 2011-000876-33 (EudraCT Number)
Record Dates: First submitted 2011-10-06; First posted 2011-10-18 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Acellular Pertussis; Hepatitis B; Haemophilus Influenzae Type b; Tetanus; Diphtheria; Poliomyelitis
MeSH Terms: conditions — Hepatitis B; Haemophilus Infections; Tetanus; Diphtheria; Poliomyelitis | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- GSK217744 Group 1 (Experimental): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation A vaccine in the primary study and a booster dose of either GSK217744 formulation A vaccine (for subjects vaccinated before Protocol Amendment 2) or Infanrix hexa vaccine (for subjects vaccinated after Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
  Interventions: Biological: Infanrix hexa; Biological: Prevenar 13; Biological: GSK217744
- GSK217744 Group 2 (Experimental): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation B vaccine in the primary study and a booster dose of either GSK217744 formulation B vaccine (for subjects vaccinated before Protocol Amendment 2) or Infanrix hexa vaccine (for subjects vaccinated after Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
  Interventions: Biological: Infanrix hexa; Biological: Prevenar 13; Biological: GSK217744
- Infanrix hexa Group (Active Comparator): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the Infanrix hexa vaccine in the primary study and a booster dose of Infanrix hexa in this study, co-administered with a booster dose of Prevenar 13. The Infanrix hexa and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
  Interventions: Biological: Infanrix hexa; Biological: Prevenar 13

INTERVENTIONS:
Biological: Infanrix hexa — Single dose, licensed formulation, intramuscular into right thigh
  Other Names: DTPa-HBV-IPV/Hib
Biological: Prevenar 13 — Single co-administered dose, intramuscular into left thigh
  Other Names: Pfizer's 13-valent pneumococcal polysaccharide conjugate vaccine
Biological: GSK217744 — Single dose, investigational formulation A or B, intramuscular into right thigh
  Arms: GSK217744 Group 1; GSK217744 Group 2

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety and reactogenicity of the booster vaccine dose of 2 new formulations of DTPa-HBV-IPV/Hib administered between 12 and 15 months of age, and the immune persistence following the primary series. All children in this booster study received a primary vaccination at 2, 3 and 4 months of age in study 113948 (NCT01248884). No new subjects will be enrolled in this booster study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the study 113948 (NCT01248884) and received three doses of the new or licensed DTPa-HBV-IPV/Hib study vaccine.
* A male or female child between, and including, 12 and 15 months of age at the time of the booster vaccination.
* Subjects who the investigator believes that parent(s)/ Legally Acceptable Representative(s) (LAR(s)) can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visit).
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period.
* Participation in another clinical study within three months prior to enrolment in the present booster study or at any time during the present booster study, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Hib vaccination or disease since the conclusion visit of study 113948 (NCT01248884).
* Serious chronic illness.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the booster dose of study vaccine or planned administration during the study period.
* Occurrence of any of the following events following previous administration of the study vaccine constitutes an absolute contraindication to further dosing.

  * Anaphylactic or other hypersensitivity reaction.
  * Encephalopathy defined as an acute, severe central nervous system disorder occurring within 7 days following vaccination and generally consisting of major alterations in consciousness, unresponsiveness, generalized or focal seizures that persist more than a few hours, with failure to recover within 24 hours.
  * Temperature of ≥ 40.0°C (axillary) or 40.5°C (rectal) within 48 hours of vaccination, not due to another identifiable cause.
  * Collapse or shock-like state (hypotonic-hyporesponsive episode) within 48 hours of vaccination.
  * Persistent, inconsolable crying occurring within 48 hours of vaccination and lasting ≥ 3 hours.
  * Seizures with or without fever occurring within 3 days of vaccination.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

• Acute disease and/or fever at the time of enrolment.

* Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting, or ≥ 38.0° on rectal setting.
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 657 (Actual)
Dates: Start 2011-10-14 (Actual); Primary Completion 2012-11-12 (Actual); Study Completion 2012-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Dominican Republic (2):
  - GSK Investigational Site, Santo Domingo
  - GSK Investigational Site, Santo Domingo, Distrito Nacional
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20051

REFERENCES:
- [Derived] Vesikari T, Rivera L, Korhonen T, Ahonen A, Cheuvart B, Hezareh M, Janssens W, Mesaros N. Immunogenicity and safety of primary and booster vaccination with 2 investigational formulations of diphtheria, tetanus and Haemophilus influenzae type b antigens in a hexavalent DTPa-HBV-IPV/Hib combination vaccine in comparison with the licensed Infanrix hexa. Hum Vaccin Immunother. 2017 Jul 3;13(7):1505-1515. doi: 10.1080/21645515.2017.1294294. Epub 2017 Mar 24. PMID 28340322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 272 subjects were enrolled in the study before the second protocol amendment and total of 385 after the amendment. After amendment 2, all subjects yet to receive a booster dose of a GSK217744 formulation, were administered the Infanrix hexa vaccine.
Period: Before Protocol Amendment 2
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Started | 85 | 88 | 99
Completed | 85 | 88 | 99
Not Completed | 0 | 0 | 0
Period: After Protocol Amendment 2.
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Started | 131 | 130 | 124
Completed | 130 | 130 | 124
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group | Total
Number analyzed (Participants) | 216 | 218 | 223 | 657
Age, Continuous [Mean (Standard Deviation); unit: Months] — Baseline measure for subjects enrolled before protocol amendment 2. Population: Data available for subjects enrolled before protocol amendment 2.
  Months
    number analyzed (Participants) | 85 | 88 | 99 | 272
    (all) | 12.9 (0.7) | 13.0 (0.7) | 13.0 (0.8) | 12.97 (0.71)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Baseline measure for subjects enrolled after protocol amendment 2. Population: Data available for subjects enrolled after protocol amendment 2.
  Months
    number analyzed (Participants) | 131 | 130 | 124 | 385
    (all) | 14.1 (0.6) | 13.9 (0.6) | 14.0 (0.6) | 14.00 (0.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measure for subjects enrolled before protocol amendment 2. Population: Data available for subjects enrolled before protocol amendment 2.
  Participants
    number analyzed (Participants) | 85 | 88 | 99 | 272
    Female | 47 | 49 | 38 | 134
    Male | 38 | 39 | 61 | 138
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measure for subjects enrolled after protocol amendment 2. Population: Data available for subjects enrolled before protocol amendment 2.
  Participants
    number analyzed (Participants) | 131 | 130 | 124 | 385
    Female | 61 | 76 | 53 | 190
    Male | 70 | 54 | 71 | 195
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Baseline measure for subjects enrolled before protocol amendment 2. Population: Data available for subjects enrolled before protocol amendment 2.
  Participants
    White - Arabic / north African heritage: number analyzed (Participants) | 85 | 88 | 99 | 272
    White - Arabic / north African heritage | 2 | 1 | 3 | 6
    White - Caucasian / European heritage: number analyzed (Participants) | 85 | 88 | 99 | 272
    White - Caucasian / European heritage | 79 | 83 | 91 | 253
    Other: Mixed: number analyzed (Participants) | 85 | 88 | 99 | 272
    Other: Mixed | 4 | 4 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Baseline measure for subjects enrolled after protocol amendment 2. Population: Data available for subjects enrolled after protocol amendment 2.
  Participants
    African heritage / African American: number analyzed (Participants) | 131 | 130 | 124 | 385
    African heritage / African American | 1 | 0 | 1 | 2
    White - Arabic / north African heritage: number analyzed (Participants) | 131 | 130 | 124 | 385
    White - Arabic / north African heritage | 0 | 0 | 3 | 3
    White - caucasian / European heritage: number analyzed (Participants) | 131 | 130 | 124 | 385
    White - caucasian / European heritage | 49 | 46 | 39 | 134
    Other: Mixed: number analyzed (Participants) | 131 | 130 | 124 | 385
    Other: Mixed | 81 | 84 | 81 | 246

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: A seroprotected subject was defined as a vaccinated subject who had anti-D and anti-T antibody concentrations ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied the booster protocol and for whom assay results were available for antibodies against at least one study vaccine antigen at the post-booster vaccination blood-sampling time point.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
Participants
  Anti-D, POST | 81 | 82 | 90
  Anti-T, POST | 81 | 82 | 90

2. Primary Outcome: Number of Seroprotected Subjects for Anti-D and Anti-T Antibodies
Description: as for outcome 1
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 118
Participants
  Anti-D, POST | 123 | 122 | 118
  Anti-T, POST | 123 | 122 | 118

3. Primary Outcome: Number of Seroprotected Subjects Against Anti-Hepatitis B (Anti-HBs) Antigens
Description: A seroprotected subject was a subject whose antibody concentration was greater than or equal to the level defining clinical protection of 10 milli-international units per millilitre (mIU/mL).
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 79 | 79 | 84
Participants | 78 | 78 | 84

4. Primary Outcome: Number of Seroprotected Subjects Against Anti-HBs Antigens
Description: as for outcome 3
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 115 | 115
Participants | 121 | 113 | 114

5. Primary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Types 1, 2 and 3
Description: A seroprotected subject was a subject whose antibody titre was greater than or equal to the level defining clinical protection of 8.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 77 | 72 | 85
Participants
  Anti-Polio 1, POST | 76 | 72 | 85
  Anti-Polio 2, POST: number analyzed (Participants) | 62 | 61 | 76
  Anti-Polio 2, POST | 62 | 60 | 76
  Anti-Polio 3, POST: number analyzed (Participants) | 64 | 63 | 73
  Anti-Polio 3, POST | 64 | 63 | 71

6. Primary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Type 1, 2 and 3
Description: as for outcome 5
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 113 | 107 | 103
Participants
  Anti-Polio 1, POST: number analyzed (Participants) | 111 | 107 | 103
  Anti-Polio 1, POST | 111 | 107 | 102
  Anti-Polio 2, POST: number analyzed (Participants) | 96 | 97 | 87
  Anti-Polio 2, POST | 96 | 96 | 87
  Anti-Polio 3, POST: number analyzed (Participants) | 113 | 103 | 98
  Anti-Polio 3, POST | 113 | 103 | 98

7. Primary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl-ribitol Phosphate (Anti-PRP)
Description: A seroprotected subject was defined as a vaccinated subject who had anti-PRP antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
Participants | 81 | 82 | 90

8. Primary Outcome: Number of Seroprotected Subjects for Anti-PRP
Description: as for outcome 7
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 118
Participants | 122 | 122 | 117

9. Primary Outcome: Concentrations for Anti-Pertussis Toxoid (Anti-PT), Anti-Filamentous Haemagglutinin (Anti-FHA), Anti-Pertactin (Anti-PRN)
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seropositivity cut-off assay was 5 EL.U/mL.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
EL.U/mL
  Anti-PT, POST: number analyzed (Participants) | 79 | 81 | 89
  Anti-PT, POST | 76.1 [66.1 to 87.6] | 74.3 [62.6 to 88.1] | 96.0 [83.5 to 110.3]
  Anti-FHA, POST | 393.7 [346.4 to 447.6] | 372.4 [332.7 to 416.7] | 423.0 [368.1 to 485.9]
  Anti-PRN, POST: number analyzed (Participants) | 81 | 81 | 89
  Anti-PRN, POST | 213.0 [178.1 to 254.7] | 180.0 [154.2 to 210.1] | 372.9 [309.3 to 449.5]

10. Primary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seropositivity cut-off assay was 5 EL.U/mL.
Time Frame: 1 month post booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 117
EL.U/mL
  Anti-PT, POST: number analyzed (Participants) | 118 | 121 | 116
  Anti-PT, POST | 92.4 [80.6 to 106.0] | 93.6 [83.1 to 105.5] | 132.6 [114.9 to 153.0]
  Anti-FHA, POST | 467.3 [417.3 to 523.3] | 446.2 [402.3 to 494.9] | 582.9 [517.1 to 657.1]
  Anti-PRN, POST: number analyzed (Participants) | 122 | 122 | 117
  Anti-PRN, POST | 253.2 [216.9 to 295.6] | 181.0 [154.8 to 211.7] | 401.1 [342.2 to 470.0]

11. Secondary Outcome: Concentrations for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.1 IU/mL.
Time Frame: Before (PRE) and 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
IU/mL
  Anti-D, POST | 5.652 [4.985 to 6.408] | 5.494 [4.891 to 6.171] | 6.772 [5.897 to 7.777]
  Anti-T, POST | 5.015 [4.341 to 5.794] | 5.034 [4.366 to 5.803] | 5.571 [4.869 to 6.374]
  Anti-D, PRE: number analyzed (Participants) | 81 | 82 | 89
  Anti-D, PRE | 0.357 [0.305 to 0.419] | 0.445 [0.381 to 0.520] | 0.401 [0.343 to 0.468]
  Anti-T, PRE: number analyzed (Participants) | 81 | 82 | 89
  Anti-T, PRE | 0.358 [0.301 to 0.427] | 0.362 [0.306 to 0.428] | 0.394 [0.337 to 0.459]

12. Secondary Outcome: Concentrations for Anti-D and Anti-T Antibodies
Description: as for outcome 11
Time Frame: Before (PRE) 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 118
IU/mL
  Anti-D, POST | 6.327 [5.698 to 7.025] | 5.452 [4.956 to 5.998] | 7.192 [6.419 to 8.059]
  Anti-T, POST | 5.986 [5.204 to 6.885] | 5.316 [4.716 to 5.992] | 5.993 [5.222 to 6.878]
  Anti-D, PRE: number analyzed (Participants) | 123 | 121 | 117
  Anti-D, PRE | 0.247 [0.213 to 0.287] | 0.278 [0.244 to 0.317] | 0.304 [0.258 to 0.360]
  Anti-T, PRE: number analyzed (Participants) | 123 | 121 | 117
  Anti-T, PRE | 0.364 [0.313 to 0.422] | 0.332 [0.289 to 0.380] | 0.331 [0.285 to 0.383]

13. Secondary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies
Description: as for outcome 1
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
Participants
  Anti-D, PRE | 78 | 80 | 84
  Anti-T, PRE | 76 | 78 | 85

14. Secondary Outcome: Number of Seroprotected Subjects for Anti-D and Anti-T Antibodies
Description: as for outcome 1
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 117
Participants
  Anti-D, PRE | 107 | 114 | 104
  Anti-T, PRE | 116 | 114 | 111

15. Secondary Outcome: Concentrations for Anti-Pertussis Toxoid (Anti-PT), Anti-Filamentous Haemagglutinin (Anti-FHA), Anti-Pertactin (Anti-PRN)
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seropositivity cut-off assay was 5 EL.U/mL.
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL.
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 89
EL.U/mL.
  Anti-PT, PRE: number analyzed (Participants) | 80 | 80 | 87
  Anti-PT, PRE | 10.5 [8.8 to 12.6] | 9.5 [7.9 to 11.4] | 12.7 [10.8 to 15.0]
  Anti-FHA, PRE: number analyzed (Participants) | 81 | 82 | 88
  Anti-FHA, PRE | 41.7 [35.4 to 49.2] | 36.9 [31.5 to 43.3] | 47.1 [40.3 to 55.1]
  Anti-PRN, PRE: number analyzed (Participants) | 81 | 81 | 89
  Anti-PRN, PRE | 12.8 [10.4 to 15.7] | 10.8 [8.9 to 13.1] | 18.2 [15.0 to 22.1]

16. Secondary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seropositivity cut-off assay was 5 EL.U/mL.
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 117
EL.U/mL
  Anti-PT, PRE | 8.3 [7.2 to 9.7] | 7.9 [6.8 to 9.1] | 9.9 [8.5 to 11.5]
  Anti-FHA, PRE: number analyzed (Participants) | 123 | 118 | 116
  Anti-FHA, PRE | 37.6 [32.5 to 43.4] | 34.0 [28.7 to 40.4] | 45.7 [38.8 to 53.9]
  Anti-PRN, PRE | 11.6 [9.7 to 13.9] | 9.7 [8.1 to 11.7] | 15.6 [13.0 to 18.7]

17. Secondary Outcome: Number of Seropositive Subjects for Anti-Pertussis Toxoid (Anti-PT), Anti-Filamentous Haemagglutinin (Anti-FHA), Anti-Pertactin (Anti-PRN)
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to (≥) the assay cut-off of 5 ELISA units per milliliter (EL.U/mL).
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
Participants
  Anti-PT, POST: number analyzed (Participants) | 79 | 81 | 89
  Anti-PT, POST | 79 | 81 | 89
  Anti-FHA, POST | 81 | 82 | 90
  Anti-PRN, POST: number analyzed (Participants) | 81 | 81 | 89
  Anti-PRN, POST | 81 | 81 | 89

18. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA, Anti-PRN
Description: as for outcome 17
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 117
Participants
  Anti-PT, POST: number analyzed (Participants) | 118 | 121 | 116
  Anti-PT, POST | 118 | 121 | 116
  Anti-FHA, POST | 123 | 122 | 117
  Anti-PRN, POST: number analyzed (Participants) | 122 | 122 | 117
  Anti-PRN, POST | 122 | 122 | 117

19. Secondary Outcome: Anti-Hepatitis B (Anti-HBs) Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seroprotection cut-off assay was 10 mIU/mL.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2))
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 79 | 79 | 84
mIU/mL | 2233.3 [1479.7 to 3370.8] | 2026.3 [1389.4 to 2955.2] | 2685.7 [1868.8 to 3859.7]

20. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seroprotection cut-off assay was 10 mIU/mL.
Time Frame: 1 month post booster vaccination (POST) ( subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 115 | 115
mIU/mL | 2229.3 [1625.5 to 3057.5] | 1729.8 [1240.6 to 2411.9] | 3711.4 [2729.7 to 5046.1]

21. Secondary Outcome: Anti-Hepatitis B (Anti-HBs) Antibody Concentration
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seroprotection cut-off assay was 10 mIU/mL.
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 74 | 79 | 84
mIU/mL | 130.3 [91.2 to 186.0] | 124.4 [89.5 to 173.0] | 166.4 [112.8 to 245.5]

22. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed as geometric mean concentrations (GMCs). Seroprotection cut-off assay was 10 mIU/mL.
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 120 | 119 | 115
mIU/mL | 94.9 [72.2 to 124.8] | 61.8 [45.7 to 83.5] | 125.9 [94.6 to 167.7]

23. Secondary Outcome: Number of Seroprotected Subjects Against Anti-Hepatitis B (Anti-HBs) Antigens
Description: as for outcome 3
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 74 | 79 | 84
Participants | 68 | 74 | 78

24. Secondary Outcome: Number of Seroprotected Subjects Against Anti-HBs Antigens
Description: as for outcome 3
Time Frame: Before (PRE) booaster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 120 | 119 | 115
Participants | 108 | 100 | 106

25. Secondary Outcome: Concentrations for Anti-poliovirus Types 1, 2, 3
Description: Concentrations were expressed as geometric mean titers (GMTs). The seroprotection cut-off of the assay was 8.
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 73 | 74 | 80
Titers
  Anti-Polio 1, PRE: number analyzed (Participants) | 69 | 74 | 71
  Anti-Polio 1, PRE | 18.2 [13.7 to 24.1] | 17.8 [13.5 to 23.5] | 22.4 [16.8 to 29.9]
  Anti-Polio 2, PRE: number analyzed (Participants) | 69 | 72 | 69
  Anti-Polio 2, PRE | 12.7 [9.5 to 16.9] | 17.1 [12.3 to 23.8] | 16.6 [12.0 to 22.8]
  Anti-Polio, 3 PRE: number analyzed (Participants) | 73 | 73 | 80
  Anti-Polio, 3 PRE | 24.7 [17.1 to 35.8] | 16.8 [12.0 to 23.5] | 26.6 [19.2 to 36.9]

26. Secondary Outcome: Concentration for Anti-poliovirus Types 1, 2, 3
Description: Concentrations were expressed as geometric mean titers (GMTs). The seroprotection cut-off of the assay was 8.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 77 | 72 | 85
Titers
  Anti-Polio 1, POST | 572.9 [435.5 to 753.6] | 558.3 [422.0 to 738.8] | 902.1 [698.4 to 1165.0]
  Anti-Polio 2, POST: number analyzed (Participants) | 62 | 61 | 76
  Anti-Polio 2, POST | 629.7 [452.6 to 876.1] | 668.7 [489.9 to 912.7] | 1184.9 [901.1 to 1558.1]
  Anti-Polio 3, POST: number analyzed (Participants) | 64 | 63 | 73
  Anti-Polio 3, POST | 1147.5 [846.2 to 1556.0] | 614.0 [453.9 to 830.6] | 1120.7 [793.0 to 1583.9]

27. Secondary Outcome: Concentrations for Anti-poliovirus Types 1, 2 and 3
Description: Concentrations were expressed as geometric mean titers (GMTs). The seroprotection cut-off of the assay was 8.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 113 | 107 | 103
Titers
  Anti-Polio 1, POST: number analyzed (Participants) | 111 | 107 | 103
  Anti-Polio 1, POST | 1121.0 [904.2 to 1389.8] | 1099.6 [905.2 to 1335.8] | 1386.2 [1091.8 to 1760.0]
  Anti-Polio 2, POST: number analyzed (Participants) | 96 | 97 | 87
  Anti-Polio 2, POST | 1485.3 [1182.4 to 1865.8] | 1215.6 [973.8 to 1517.4] | 1537.2 [1191.0 to 1984.1]
  Anti-Polio 3, POST: number analyzed (Participants) | 113 | 103 | 98
  Anti-Polio 3, POST | 1851.2 [1473.2 to 2326.1] | 1960.4 [1574.0 to 2441.5] | 2376.4 [1874.2 to 3013.2]

28. Secondary Outcome: Concentration for Anti-poliovirus Type 1, 2 and 3
Description: Concentrations were expressed as geometric mean titers (GMTs). The seroprotection cut-off of the assay was 8.
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 108 | 109 | 104
Titers
  Anti-Polio 1, PRE: number analyzed (Participants) | 106 | 105 | 99
  Anti-Polio 1, PRE | 53.5 [39.6 to 72.4] | 50.7 [37.2 to 69.2] | 70.8 [52.4 to 95.8]
  Anti-Polio 2, PRE: number analyzed (Participants) | 90 | 93 | 85
  Anti-Polio 2, PRE | 76.6 [50.3 to 116.7] | 55.0 [38.2 to 79.3] | 82.7 [55.6 to 122.9]
  Anti-Polio, 3 PRE | 67.8 [47.3 to 97.2] | 73.8 [52.2 to 104.2] | 93.9 [64.4 to 136.8]

29. Secondary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Type 1, 2 and 3
Description: as for outcome 5
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 73 | 74 | 80
Participants
  Anti-Polio 1, PRE: number analyzed (Participants) | 69 | 74 | 71
  Anti-Polio 1, PRE | 50 | 54 | 56
  Anti-Polio 2, PRE: number analyzed (Participants) | 69 | 72 | 69
  Anti-Polio 2, PRE | 38 | 44 | 44
  Anti-Polio, 3 PRE: number analyzed (Participants) | 73 | 73 | 80
  Anti-Polio, 3 PRE | 51 | 43 | 61

30. Secondary Outcome: Number of Seroprotected Subjects Against Anti-Poliovirus Type 1, 2 and 3
Description: as for outcome 5
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 108 | 109 | 104
Participants
  Anti-Polio 1, PRE: number analyzed (Participants) | 106 | 105 | 99
  Anti-Polio 1, PRE | 95 | 91 | 92
  Anti-Polio 2, PRE: number analyzed (Participants) | 90 | 93 | 85
  Anti-Polio 2, PRE | 78 | 81 | 74
  Anti-Polio, 3 PRE | 96 | 99 | 91

31. Secondary Outcome: Concentrations for Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibodies
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seroprotection cut-off of the assay was 0.15 µg /mL.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 90
µg /mL | 12.765 [9.300 to 17.520] | 15.904 [11.723 to 21.576] | 17.099 [12.966 to 22.550]

32. Secondary Outcome: Concentrations for Anti-PRP Antibodies
Description: as for outcome 31
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 122 | 118
µg /mL | 21.462 [16.650 to 27.664] | 15.903 [12.132 to 20.848] | 17.429 [13.429 to 22.620]

33. Secondary Outcome: Concentrations for Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibodies
Description: as for outcome 31
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 89
µg /mL | 0.173 [0.138 to 0.216] | 0.175 [0.142 to 0.216] | 0.236 [0.182 to 0.307]

34. Secondary Outcome: Concentrations for Anti-polyribosyl-ribitol Phosphate Antibodies
Description: as for outcome 31
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2))
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 117
µg /mL | 0.328 [0.262 to 0.409] | 0.288 [0.227 to 0.365] | 0.334 [0.254 to 0.439]

35. Secondary Outcome: Number of Seropositive Subjects for Anti-Pertussis Toxoid (Anti-PT), Anti-Filamentous Haemagglutinin (Anti-FHA), Anti-Pertactin (Anti-PRN)
Description: as for outcome 17
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 89
Participants
  Anti-PT, PRE: number analyzed (Participants) | 80 | 80 | 87
  Anti-PT, PRE | 68 | 65 | 78
  Anti-FHA, PRE: number analyzed (Participants) | 81 | 82 | 88
  Anti-FHA, PRE | 81 | 81 | 88
  Anti-PRN, PRE: number analyzed (Participants) | 81 | 81 | 89
  Anti-PRN, PRE | 68 | 69 | 83

36. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA, Anti-PRN
Description: as for outcome 17
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 117
Participants
  Anti-PT, PRE | 95 | 94 | 97
  Anti-FHA, PRE: number analyzed (Participants) | 123 | 118 | 116
  Anti-FHA, PRE | 122 | 117 | 116
  Anti-PRN, PRE | 98 | 92 | 105

37. Secondary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl-ribitol Phosphate (Anti-PRP)
Description: as for outcome 7
Time Frame: Before (PRE) booster vaccination (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 89
Participants | 41 | 45 | 52

38. Secondary Outcome: Number of Seroprotected Subjects for Anti-PRP
Description: as for outcome 7
Time Frame: Before (PRE) booster vaccination (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 117
Participants | 92 | 78 | 81

39. Secondary Outcome: Concentrations for Anti-pneumococcal (Anti-PNE) Antibodies
Description: Concentrations were expressed as geometric mean concentrations (GMCs). The seropositivity cut-off of the assay was 0.15 µg /mL. The anti-PNE serotypes assessed were 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 50 | 50 | 53
µg /mL
  Anti- PNE 1 | 2.07 [1.69 to 2.53] | 2.16 [1.75 to 2.68] | 2.27 [1.84 to 2.80]
  Anti- PNE 3: number analyzed (Participants) | 40 | 44 | 44
  Anti- PNE 3 | 0.76 [0.62 to 0.93] | 0.87 [0.66 to 1.15] | 0.88 [0.69 to 1.14]
  Anti- PNE 4 | 1.87 [1.51 to 2.32] | 1.83 [1.46 to 2.28] | 2.14 [1.72 to 2.66]
  Anti- PNE 5 | 1.18 [0.97 to 1.42] | 1.10 [0.92 to 1.33] | 1.21 [0.99 to 1.49]
  Anti- PNE 6A | 7.71 [6.49 to 9.16] | 6.92 [5.53 to 8.64] | 8.63 [6.79 to 10.96]
  Anti- PNE 6B | 4.24 [3.39 to 5.30] | 4.21 [3.17 to 5.59] | 4.58 [3.45 to 6.08]
  Anti- PNE 7F | 3.27 [2.75 to 3.89] | 3.42 [2.94 to 3.97] | 4.27 [3.58 to 5.08]
  Anti- PNE 9V | 1.68 [1.33 to 2.11] | 1.52 [1.25 to 1.85] | 1.63 [1.29 to 2.06]
  Anti- PNE 14 | 8.22 [6.27 to 10.77] | 8.80 [7.01 to 11.06] | 8.97 [7.29 to 11.02]
  Anti- PNE 18C | 1.50 [1.13 to 1.99] | 1.63 [1.32 to 2.01] | 1.64 [1.33 to 2.02]
  Anti- PNE 19A: number analyzed (Participants) | 49 | 50 | 53
  Anti- PNE 19A | 7.00 [5.76 to 8.51] | 8.05 [6.39 to 10.13] | 6.70 [5.14 to 8.73]
  Anti- PNE 19F | 7.15 [5.86 to 8.74] | 7.34 [5.89 to 9.15] | 6.72 [5.32 to 8.48]
  Anti- PNE 23F: number analyzed (Participants) | 50 | 47 | 52
  Anti- PNE 23F | 3.74 [2.87 to 4.88] | 4.54 [3.67 to 5.63] | 3.94 [2.97 to 5.23]

40. Secondary Outcome: Concentrations for Anti-PNE Antibodies
Description: as for outcome 39
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg /mL
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 23 | 21 | 20
µg /mL
  Anti- PNE 1 | 2.54 [1.93 to 3.34] | 2.47 [1.83 to 3.35] | 3.47 [2.23 to 5.41]
  Anti- PNE 3: number analyzed (Participants) | 21 | 18 | 16
  Anti- PNE 3 | 0.76 [0.59 to 0.96] | 0.82 [0.60 to 1.13] | 0.92 [0.66 to 1.30]
  Anti-PNE 4 | 2.03 [1.53 to 2.68] | 2.10 [1.59 to 2.79] | 2.57 [1.65 to 4.01]
  Anti-PNE 5 | 1.26 [0.97 to 1.63] | 1.24 [0.98 to 1.57] | 1.29 [0.89 to 1.87]
  Anti-PNE 6A | 10.64 [7.94 to 14.25] | 7.67 [6.18 to 9.53] | 7.47 [4.76 to 11.70]
  Anti-PNE 6B | 5.04 [3.74 to 6.79] | 4.56 [3.16 to 6.59] | 6.62 [3.90 to 11.24]
  Anti-PNE 7F | 4.20 [3.45 to 5.11] | 3.97 [2.98 to 5.29] | 4.67 [3.16 to 6.89]
  Anti-PNE 9V | 2.20 [1.66 to 2.93] | 1.42 [1.10 to 1.85] | 1.85 [1.21 to 2.83]
  Anti-PNE 14 | 7.47 [5.68 to 9.83] | 8.12 [6.04 to 10.93] | 9.28 [6.15 to 14.01]
  Anti-PNE 18C | 1.80 [1.34 to 2.40] | 1.52 [1.09 to 2.11] | 2.09 [1.41 to 3.11]
  Anti-PNE 19A | 8.79 [6.53 to 11.82] | 6.22 [4.99 to 7.76] | 9.10 [5.23 to 15.84]
  Anti-PNE 19F | 8.09 [5.48 to 11.95] | 7.11 [5.21 to 9.70] | 5.56 [3.38 to 9.14]
  Anti-PNE 23F | 5.31 [4.29 to 6.57] | 4.00 [3.05 to 5.24] | 5.82 [3.59 to 9.44]

41. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal (Anti-PNE) Serotypes
Description: A seropositive subject was defined as a vaccinated subject who had anti- pneumococcal antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL). The anti-PNE serotypes assessed were 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 50 | 50 | 53
Participants
  Anti- PNE 1 | 50 | 50 | 53
  Anti- PNE 3: number analyzed (Participants) | 40 | 44 | 44
  Anti- PNE 3 | 40 | 43 | 43
  Anti- PNE 4 | 50 | 50 | 53
  Anti- PNE 5 | 50 | 50 | 53
  Anti- PNE 6A | 50 | 50 | 53
  Anti- PNE 6B | 50 | 49 | 53
  Anti- PNE 7F | 50 | 50 | 53
  Anti- PNE 9V | 50 | 50 | 53
  Anti- PNE 14 | 49 | 50 | 53
  Anti- PNE 18C | 49 | 50 | 53
  Anti- PNE 19A: number analyzed (Participants) | 49 | 50 | 53
  Anti- PNE 19A | 49 | 50 | 53
  Anti- PNE 19F | 50 | 50 | 53
  Anti- PNE 23F: number analyzed (Participants) | 50 | 47 | 52
  Anti- PNE 23F | 50 | 47 | 52

42. Secondary Outcome: Number of Seropositive Subjects for Anti-PNE Serotypes
Description: as for outcome 41
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 23 | 21 | 20
Participants
  Anti- PNE 1 | 23 | 21 | 20
  Anti- PNE 3: number analyzed (Participants) | 21 | 18 | 16
  Anti- PNE 3 | 21 | 18 | 16
  Anti-PNE 4 | 23 | 21 | 20
  Anti-PNE 5 | 23 | 21 | 20
  Anti-PNE 6A | 23 | 21 | 20
  Anti-PNE 6B | 23 | 21 | 20
  Anti-PNE 7F | 23 | 21 | 20
  Anti-PNE 9V | 23 | 21 | 20
  Anti-PNE 14 | 23 | 21 | 20
  Anti-PNE 18C | 23 | 21 | 20
  Anti-PNE 19A: number analyzed (Participants) | 23 | 21 | 19
  Anti-PNE 19A | 23 | 21 | 19
  Anti-PNE 19F | 23 | 21 | 20
  Anti-PNE 23F | 23 | 21 | 20

43. Secondary Outcome: Number of Subjects With Booster Response to Anti-pertussis Antigens (Anti-PT, Anti-FHA and Anti-PRN)
Description: Booster response defined as : - For initially seronegative subjects, antibody concentration ≥ 5 EL.U/mL one month after booster vaccination - For initially seropositive subjects, antibody concentration at Post-booster ≥ 2 fold the pre-vaccination antibody concentration
Time Frame: 1 month post booster vaccination (POST) (subjects enrolled before protocol amendment 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 81 | 82 | 88
Participants
  Anti-PT: number analyzed (Participants) | 78 | 79 | 86
  Anti-PT | 72 | 77 | 86
  Anti-FHA | 79 | 81 | 87
  Anti-PRN: number analyzed (Participants) | 81 | 80 | 88
  Anti-PRN | 81 | 80 | 87

44. Secondary Outcome: Number of Subjects With Booster Response to Anti-pertussis Antigens
Description: as for outcome 43
Time Frame: 1 month poste booster vaccination (POST) (subjects enrolled after protocol amendment 2)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 123 | 121 | 116
Subjects
  Anti-PT: number analyzed (Participants) | 118 | 121 | 115
  Anti-PT | 118 | 119 | 110
  Anti-FHA: number analyzed (Participants) | 123 | 118 | 115
  Anti-FHA | 120 | 115 | 113
  Anti-PRN: number analyzed (Participants) | 122 | 121 | 116
  Anti-PRN | 121 | 120 | 115

45. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period. (subjects enrolled before protocol amendment 2)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 85 | 88 | 99
Participants
  Any pain | 56 | 67 | 63
  Any redness | 55 | 56 | 59
  Any swelling | 45 | 43 | 48

46. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptom
Description: as for outcome 45
Time Frame: During the 4-day (Days 0-3) post-vaccination period. (subjects enrolled after protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 131 | 130 | 124
Participants
  Any pain | 76 | 66 | 64
  Any redness | 47 | 36 | 40
  Any swelling | 43 | 34 | 38

47. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited local symptoms assessed were drowsiness, irritability/fussiness, loss of appetite and fever [axillary temperature above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period. (subjects enrolled before protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 85 | 88 | 99
Participants
  Any drowsiness | 54 | 47 | 47
  Any irritability/fussiness | 69 | 73 | 74
  Any loss of appetite | 43 | 45 | 46
  Any fever | 42 | 41 | 37

48. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptom
Description: as for outcome 47
Time Frame: During the 4-day (Days 0-3) post-vaccination period. (subjects enrolled after protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 131 | 130 | 124
Participants
  Any drowsiness | 52 | 40 | 40
  Any irritability/fussiness | 66 | 58 | 62
  Any loss of appetite | 42 | 37 | 34
  Any fever | 58 | 50 | 52

49. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an AE regardless of intensity grade or relationship to study vaccination.
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination. (subjects enrolled before protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 85 | 88 | 99
Participants | 42 | 39 | 67

50. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: as for outcome 49
Time Frame: Within the 31-day (Days 0-30) follow up period after vaccination. (subjects enrolled after protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 131 | 130 | 124
Participants | 38 | 27 | 31

51. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Any SAE = any SAE regardless of assessment of relationship to study vaccination.
Time Frame: During the entire study period (Days 0-30). (subjects enrolled before protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 85 | 88 | 99
Participants | 0 | 0 | 0

52. Secondary Outcome: Number of Subjects Reporting Any SAEs
Description: as for outcome 51
Time Frame: During the entire study period (Days 0-30). (subjects enrolled after protocol amendment 2)
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | GSK217744 Group 1 | GSK217744 Group 2 | Infanrix Hexa Group
Number analyzed (Participants) | 131 | 130 | 124
Participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: 4-day follow-up period after vaccination; unsolicited AEs: 31-day follow-up period after vaccination; SAEs: during the entire study period (Days 0-30).
Groups:
- GSK217744 Group 1(Before Protocol Amendment2): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation A vaccine in the primary study and a booster dose of GSK217744 formulation A vaccine (for subjects vaccinated before Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
- GSK217744 Group 2(Before Protocol Amendment2): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation B vaccine in the primary study and a booster dose of GSK217744 formulation B vaccine (for subjects vaccinated before Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
- Infanrix Hexa Group(Before Protocol Amendment2); Infanrix Hexa Group(After Protocol Amendment2): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the Infanrix hexa vaccine in the primary study and a booster dose of Infanrix hexa in this study, co-administered with a booster dose of Prevenar 13. The Infanrix hexa and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
- GSK217744 Group 1(After Protocol Amendment2): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation A vaccine in the primary study and a booster dose of Infanrix hexa vaccine (for subjects vaccinated after Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
- GSK217744 Group 2(After Protocol Amendment2): Subjects aged between and including 12 and 15 months at the time of booster vaccination who received the GSK217744 formulation B vaccine in the primary study and a booster dose of Infanrix hexa vaccine (for subjects vaccinated after Protocol Amendment 2) in this study, coadministered with a booster dose of Prevenar 13. The Infanrix hexa/GSK217744 and Prevenar 13 vaccines were administered intramuscularly into the right and left sides of the thigh, respectively.
Arm/Group | GSK217744 Group 1(Before Protocol Amendment2) | GSK217744 Group 2(Before Protocol Amendment2) | Infanrix Hexa Group(Before Protocol Amendment2) | GSK217744 Group 1(After Protocol Amendment2) | GSK217744 Group 2(After Protocol Amendment2) | Infanrix Hexa Group(After Protocol Amendment2)
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/88 | 0/99 | 0/131 | 0/130 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/88 | 0/99 | 0/131 | 2/130 | 0/124
Other Adverse Events (participants affected / at risk) | 85/85 | 85/88 | 96/99 | 118/131 | 103/130 | 104/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK217744 Group 1(Before Protocol Amendment2) (N=85) | GSK217744 Group 2(Before Protocol Amendment2) (N=88) | Infanrix Hexa Group(Before Protocol Amendment2) (N=99) | GSK217744 Group 1(After Protocol Amendment2) (N=131) | GSK217744 Group 2(After Protocol Amendment2) (N=130) | Infanrix Hexa Group(After Protocol Amendment2) (N=124)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK217744 Group 1(Before Protocol Amendment2) (N=85) | GSK217744 Group 2(Before Protocol Amendment2) (N=88) | Infanrix Hexa Group(Before Protocol Amendment2) (N=99) | GSK217744 Group 1(After Protocol Amendment2) (N=131) | GSK217744 Group 2(After Protocol Amendment2) (N=130) | Infanrix Hexa Group(After Protocol Amendment2) (N=124)
Conjunctivitis (Infections and infestations) | 3 | 1 | 7 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 4 | 2 | 2 | 4
Injection site induration (General disorders) | 7 | 3 | 5 | 4 | 0 | 0
Pyrexia (General disorders) | 44 | 45 | 39 | 59 | 51 | 52
Pain (General disorders) | 56 | 67 | 63 | 76 | 66 | 64
Erythema (Skin and subcutaneous tissue disorders) | 55 | 56 | 59 | 47 | 36 | 40
Swelling (General disorders) | 45 | 43 | 48 | 43 | 34 | 38
Somnolence (Nervous system disorders) | 54 | 47 | 47 | 52 | 40 | 40
Decreased appetite (Metabolism and nutrition disorders) | 43 | 45 | 46 | 42 | 37 | 34
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5 | 13 | 9 | 8
Otitis media (Infections and infestations) | 6 | 11 | 11 | 3 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 9 | 1 | 1 | 4
Gastroenteritis (Infections and infestations) | 2 | 2 | 5 | 1 | 1 | 1
Irritability (Psychiatric disorders) | 69 | 73 | 74 | 66 | 58 | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.